CLINICAL TRIAL: NCT06640569
Title: Preliminary Characterization of Commercial Kratom Extract Products
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00440647
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Kratom Pharmacodynamics; Kratom Pharmacokinetics
Keywords: kratom; kratom extracts; pharmacokinetics; behavioral pharmacology; Mitragyna speciosa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma; urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- US Adult Kratom Extract Consumers: Participants who regularly consume commercial kratom extracts will orally self-administer a single serving of their commercial kratom extract product under direct observation in order to evaluate acute physiological, subjective, and cognitive effects and determine pharmacokinetics. Participants will undergo direct observation and assessment for acute self-administration and for a period following the peak effects (i.e., a period of short abstinence). Physiological, subjective, and cognitive effects will be measured in an inpatient unit where the participant will reside for 2 days and 1 night (consecutive).

SUMMARY:
To understand the acute subjective, physiological, and cognitive effects of commercial kratom extract products among US adults who consume these products regularly, and to understand how these products are metabolized by the human body.

DETAILED DESCRIPTION:
Kratom products, made from the botanical Mitragyna speciosa, have proliferated in the United States since 2006 and now include a variety of brands and formulations. Kratom whole-leaf products and kratom leaf-derived extract products are the two major types of products within the marketplace. To date, most studies have examined kratom whole-leaf products, both in terms of self-report from consumers and in terms of two US-based, small lab-based pharmacokinetic/pharmacodynamic (PK/PD) studies. In order to follow-up on the investigators' prior work examining the acute effects of kratom in adults (age 21 or older) who regularly use whole-leaf kratom products, the investigators propose a pilot study (N=16) that purposefully samples US adults who use popular kratom extract products sold legally in most of US, including the state of Maryland. Despite the widespread use of kratom extract products, particularly among the best-selling brands, the investigators have no independently collected and published data derived from human laboratory studies on the PK/PD associated with these products. The investigators will conduct a within-person, single-dose pilot study wherein 16 adult consumers of kratom extract products will self-administer a single oral dose of the participant's kratom extract. As this is an exploratory pilot study, the investigators are not making a priori hypothesis. Rather, this is a proof-of-concept pilot study needed to first measure the basic PK and PD (physiological, subjective, cognitive) responses to extract product servings taken by adults who consumed the extracts regularly. There is immediate public health need to better understand kratom extract consumer experiences given that these products are unregulated but widely used. Such data have ecological validity and can inform next steps for funding and research.

ELIGIBILITY:
Inclusion Criteria:

* 1) >21 years old;
* 2) Experienced kratom extract product consumer of one of the leading US brands listed in the study protocol;
* 3) Reports a specific kratom extract product brand and specific dose amount (or range of typical dose amount) on the online screener;
* 4) English language proficient;
* 5) Willingness to provide requested samples of the kratom extract product currently being taken.

Exclusion Criteria:

* 1) Reports any acute adverse or unexpected or otherwise sudden health event related to their typical kratom product dose that occurred within 30 days of screening;
* 2) Having ever sought medical attention for an acute adverse health event as a result of taking any kratom product;
* 3) Cannot or will not provide their kratom extract product samples in the form of an unopened package that is clearly labeled with at least the product and vendor name;
* 4)The kratom extract product used by the participant has any semi-synthetic or fully synthetic ingredient listed or is known by the study team to have such an ingredient;
* 5) Currently breastfeeding or pregnant;
* 6) history or current diagnosis of psychotic disorder;
* 7) current untreated bipolar disorder; 8) current untreated major depressive disorder;
* 8) Current physical dependence on alcohol, benzodiazepines, or opioids (self-reported or otherwise evidenced) requiring medical intervention;
* 9) Reports use of fentanyl within the past month and/or has a fentanyl positive drug screen;
* 10) Discordance between self-reported substance use and drug screen results obtained during screening;
* 11)Any physical, psychiatric, environmental, situational, or kratom product-related condition considered by the study team to increase risk or undue burden.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: US adults who use kratom extract products on a regular basis
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-11-11 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Drug Effects Questionnaire | Administered at 7 timepoints on Study Days 1-2
  Drug Effects Questionnaire (DEQ) visual analogue scale (0-100) rating for DEQ item "feeling" effects and "liking" effects. 0 is the measure of least impactful 'effect'.
Cognitive Effects as assessed by the Digit Symbol Substitution Task | Administered at 7 time points on Study Days 1-2
  The 2-minute computerized Digit Symbol Substitution Task (DSST) outcome of total number of correct responses (accuracy) within the 2-minute test window. This will evaluate cognitive performance and impairment.
Pupil size | Measured at 7 timepoints on Study Days 1-2
  Pupil diameter in mm under stable light conditions using a pupilometer.
Resting Heart Rate | Measured at 7 timepoints on Study Days 1-2
  Resting heart rate in beats per minute.

SECONDARY OUTCOMES:
Qualitative Interview | Study Day 2
  Qualitative interview of participants' experience with kratom products and how use has changed over time. Will take approximately 1.5 - 2 hours to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten E Smith, MSW, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University Behavioral Pharmacology Research Unit, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Data sharing agreements/materials will be implemented to share biospecimen data and limited datasets with deidentified participant information to collaborators for bioanalytics. No protected health information or personally identifiable information will be shared and all data will be coded with unique participant Identification.
Supporting Information: Study Protocol, ICF
Time Frame: After the study has concluded or upon request.
Access Criteria: Researchers and scientists university/academic or government settings (non-commercial, non-industry settings) can make a request to the PI.